CLINICAL TRIAL: NCT02764554
Title: Post-Marketing Surveillance of Lenvima in Korean Patients
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E7080-M065-502
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2021-10-07 (Actual); Status verified 2021-08

CONDITIONS: Differentiated Thyroid Carcinoma (DTC)
Keywords: Post-Marketing Surveillance; Lenvima; Lenvatinib; E7080; Differentiated thyroid carcinoma; Refractory to radioactive iodine; Progressive; locally recurrent; metastatic
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lenvatinib 4 milligram (mg) and 10 mg capsule: Participants who are prescribed with Lenvatinib per approved prescribing information of lenvatinib in normal clinical practice setting.

SUMMARY:
The purpose of this post-marketing surveillance (PMS) is to observe the safety profile of Lenvima (lenvatinib) in normal clinical practice setting.

ELIGIBILITY:
Inclusion criteria:

Participants who meet the following criteria will be eligible for inclusion in the study:

1. Participants with approved indication for lenvatinib in Korea
2. Participants who have written consent for use of personal and medical information for the study purpose

Exclusion Criteria:

Investigators will refer to approved indications and contraindications regarding exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who are prescribed with Lenvatinib per approved prescribing information of lenvatinib in normal clinical practice setting.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events, Serious Adverse Events, and Adverse Drug Reactions | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (32):
- South Korea (32):
  - Eisai Trial Site #18, Anyang, Gyeongji-do
  - Eisai Trial Site #30, Bundang, Gyeongji-do
  - Eisai Trial Site #14, Goyang, Gyeongji-do
  - Eisai Trial Site #27, Goyang, Gyeongji-do
  - Eisai Trial Site #34, Goyang, Gyeongji-do
  - Eisai Trial Site #21, Suwon, Gyeongji-do
  - Eisai Trial Site #24, Yangsan, Gyeongsangnam-do
  - Eisai Trial Site #15, Busan
  - Eisai Trial Site #16, Busan
  - Eisai Trial Site #17, Busan
  - Eisai Trial Site #20, Busan
  - Eisai Trial Site #22, Busan
  - Eisai Trial Site #37, Busan
  - Eisai Trial Site #36, Daegu
  - Eisai Trial Site #4, Daegu
  - Eisai Trial Site #13, Gwangju
  - Eisai Trial Site #25, Incheon
  - Eisai Trial Site #26, Incheon
  - Eisai Trial Site #32, Incheon
  - Eisai Trial Site #19, Jeju City
  - Eisai Trial Site #1, Seoul
  - Eisai Trial Site #23, Seoul
  - Eisai Trial Site #29, Seoul
  - Eisai Trial Site #31, Seoul
  - Eisai Trial Site #33, Seoul
  - Eisai Trial Site #35, Seoul
  - Eisai Trial Site #38, Seoul
  - Eisai Trial Site #39, Seoul
  - Eisai Trial Site #8, Seoul
  - Eisai Trial Site #9, Seoul
  - Eisai Trial Site #12, Ulsan
  - Eisai Trial Site #6, Ulsan